CLINICAL TRIAL: NCT03246412
Title: Nevus or Melanoma? Nevus Doctor - Computer Aided Clinical Decision Support in Primary Health Care
Brief Title: Nevus Doctor Clinical Decision Support for GPs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of North Norway (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2013/1793
Record Dates: First submitted 2017-08-08; First posted 2017-08-11 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Melanoma (Skin); Non-melanoma Skin Cancer; Actinic Keratoses
MeSH Terms: conditions — Melanoma; Keratosis, Actinic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nevus doctor clinical decision support (Experimental): The GPs have access to the clinical decision support tool "Nevus doctor".
  Interventions: Diagnostic Test: Nevus doctor clinical decision support
- Control (No Intervention): The GPs have no access to the clinical decision support tool "Nevus Doctor".

INTERVENTIONS:
Diagnostic Test: Nevus doctor clinical decision support — The computer program analyzes dermatoscopic images. The output is an estimate of the risk of the skin lesion representing skin cancer. The decision support tool helps the doctor to assess the significance of the computer output by taking into account clinical information.
  Arms: Nevus doctor clinical decision support

SUMMARY:
The study investigates if a computer-based clinical decision support tool for skin cancer may improve the diagnostic accuracy of general practitioners (GPs). The aim of the program is to help GPs increase their diagnostic accuracy, in particular regarding the selection of suspicious skin lesions that need biopsy or referral to specialist health care for further assessment. Half of the physicians in the trial will have the clinical decision support tool available during consultations, while the other half has no such tool available. We hypothesize that general practitioners using the clinical decision support tool will have a higher number of correct classifications of skin lesions compared to doctors without the tool.

DETAILED DESCRIPTION:
General practitioners (GPs) examine patients who attend a primary health care center. In the intervention group the computer-based clinical decision support tool "Nevus doctor" in a first step assists doctors in the process of selecting skin lesions that are suggestive of cancer. In the next step a given skin lesion is photographed using a dermatoscope attached to the lens of the camera. The dermatoscopic image is then processed by the computer program "Nevus doctor" and a preliminary result is presented. Finally the GP reviews the result and assesses the clinical significance of the output by using guidelines presented by "Nevus doctor". The patient is subsequently referred to a dermatologist and a complete skin examination is performed. The assessment of the dermatologist serves as the gold standard.

ELIGIBILITY:
Inclusion Criteria:

* Patients concerned about one or several skin lesion(s)
* Patients with any other condition if doctor has observed a skin lesion suspicious for skin cancer (incl. actinic keratosis)

Exclusion Criteria:

* Patients not able to give consent

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2018-01-17 (Actual); Primary Completion 2019-12-12 (Actual); Study Completion 2019-12-12 (Actual)

PRIMARY OUTCOMES:
Diagnostic classification of suspicious skin lesions | Up to 3 months
  Skin lesions selected by the GP are classified into three classes: 1 Not suspicious for skin cancer, 2 Somewhat suspicious for skin cancer, 3 Very suspicious for skin cancer. The reference standard is the specialist's classification. The number of correct classifications are counted. Sensitivity and specificity scores are calculated.

SECONDARY OUTCOMES:
Skin lesions not classified by GPs | Up to 3 months
  Skin lesions that were not selected by the GP but were later classified by the specialist to be suspicious for skin cancer or very suspicious for skin cancer are counted.
Biopsies and excisions | Up to 3 months
  Skin lesions biopsied or excised by the GP are counted.

OTHER OUTCOMES:
User experience | Up to 12 months.
  The GPs are asked to answer a questionnaire to assess the user experiences of operating the clinical decision support tool.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Schopf, PhD, Principal Investigator — University Hospital of North Norway
Locations (1):
- University Hospital of North-Norway, Tromsø, Troms, Norway

IPD SHARING:
Plan to Share IPD: No